CLINICAL TRIAL: NCT04193254
Title: Relation of Pulmonary Protective Ventilation, Mechanical Power and Driving Pressure With Mortality and SOFA of Mechanically Ventilated Patients in ER, Ward and ICU at General Hospital 11 IMSS Piedras Negras, Coahuila
Brief Title: LPP , MP and DP:Relation With Mortality and SOFA in Mechanically Ventilated Patients in ER, Ward and ICU
Acronym: LUMEDRI-MORT
Status: Completed | Type: Observational
Sponsor: JOSE IVAN RODRIGUEZ DE MOLINA SERRANO (Other)
Responsible Party: Sponsor-Investigator, JOSE IVAN RODRIGUEZ DE MOLINA SERRANO, Head of ICU Jose Ivan RodriguezdeMolina Critical Care Ph., IMSS Hospital General de Zona 11, Piedras Negras
Organization: IMSS Hospital General de Zona 11, Piedras Negras (Other)
Other Study IDs: R-2019-506-010
Record Dates: First submitted 2019-08-23; First posted 2019-12-10 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Mechanical Ventilation Complication; Mechanical Power; Driving Pressure; Lung Protective Ventilation
Keywords: lung protective ventilation; mechanical power; driving pressure; SOFA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational, longitudinal study, September 2019 to March 2020 of all adult patients who required invasive mechanical ventilation treated at General Hospital of Zone 11 IMSS in Piedras Negras, Coahuila. The investigators aim to assess the relation of lung protective ventilation, mechanical power and driving pressure in mortality and SOFA of mechanically ventilated patients inside and outside ICU at the General Hospital of Zona 11 Piedras Negras, IMSS

DETAILED DESCRIPTION:
Prospective, observational, longitudinal study from Sept 2019 to Feb 2020 of all adult patients who required invasive mechanical ventilation treated at General Hospital of Zone 11 IMSS in Piedras Negras Coahuila.

Independent variable: Lung protective ventilation, Mechanical power, Driving pressure Dependent variable: Hospital Mortality, Sequential Organic Failure Assessment (SOFA)

Also will be registered:

1. Primary diagnosis
2. Compliance with lung protective ventilation
3. Complications associated to mechanical ventilation
4. Quality of attention indicators for MV patients as defined by Semicyuc.
5. Real mortality vs Expected mortality analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years or older, with invasive mechanical ventilation

Exclusion Criteria:

* Patients with 17 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that required invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation of Lung protective ventilation with mortality and SOFA (Sequential Organic Failure Assessment) | Sept 19-Feb 20
  Lung Protective Ventilation: Qualitative variable will be defined as YES or NO with the averages of the daily measurements of tidal volume and Pressure plateau. It is defined as Tidal volume (Vc or Vt) <8 ml / kg (ideal weight) and Plateau or plateau pressure (Ppl, Pm) <30cmH2O
Correlation of mechanical power with mortality and SOFA | Sept 19-Feb 20
  Mechanical power: Quantitative variable. calculated using Marinni equation: MP= (0.098)x(Plateau pressure-PEEP)x Respiratory Rate xTidal Volume. Normal range < 13
Correlation of driving pressure with mortality and SOFA | Sept 19-Feb 20
  Driving Pressure: Quantitative variabel, calculated using: Pplateau pressure-PEEP. nomral range < 13

CONTACTS AND LOCATIONS:
Overall Officials: JOSE IVAN RODRIGUEZ DE MOLINA SERRANO, MD, Principal Investigator — HGZ 11 IMSS PIEDRAS NEGRAS COAHUILA
Locations (1):
- Hospital General Zona 11 Imss Piedras Negras Coahuila, Piedras Negras, Coahuila, Mexico